CLINICAL TRIAL: NCT06927856
Title: Test-to-PrEP: A Randomized Hybrid Implementation/Effectiveness Trial of a Social Network Strategy to Increase Equitable Reach of HIV Testing and PrEP Information
Brief Title: The Test-to-PrEP Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susanne Doblecki-Lewis, Professor of Clinical Medicine, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20240478; R01MH138190-01 (NIH)
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test-to-PrEP group (Experimental): Participants in this group will receive the Test-to-PrEP intervention for up to 1 year
  Interventions: Behavioral: Test-to-PrEP
- Access by Referral group (Experimental): Participants in this group will receive the Access by Referral intervention for up to 1 year
  Interventions: Behavioral: Access by Referral

INTERVENTIONS:
Behavioral: Test-to-PrEP — Participants, called Egos, will come once to the clinic throughout the duration of the study, for up to 1 hour. During the visit, participants will receive up to 4 Test-to-PrEP Packs, which include an HIV self-test kit and HIV prevention education materials and a brief (approximately 15 minutes) training. The training includes instructions on how to initiate conversations related to HIV, HIV testing, and HIV prevention, as well as proper handling of the HIV self-test kit. Participants are asked to distribute the Test-to-PrEP Packs to Social Network Contacts (peers), called Alters.
  Arms: Test-to-PrEP group
Behavioral: Access by Referral — Participants, called Egos, will receive up to 4 Access by Referral Cards once. Participants will receive a brief (approximately 15 minutes) training. The training includes instructions on how to initiate conversations related to HIV, HIV testing, and HIV prevention, as well as proper handling of the HIV self-test kit. Participants are asked to distribute the Access by Referral Cards to Social Network Contacts (peers), also called Alters. The Referral Card can be used to order a Test-to-PrEP Pack, including the HIV self-test and HIV prevention education material, that will be mailed to an address of the Alter's choice.
  Arms: Access by Referral group

SUMMARY:
To compare the effectiveness of two social network strategies (direct distribution and referral-based distribution) in increasing HIV self-testing (HIVST) completion rates among social network contacts of current Pre-Exposure Prophylaxis (PrEP) clients.

ELIGIBILITY:
Inclusion Criteria - PrEP Clients (Egos):

* Stated willingness to provide informed consent.
* Stated willingness to comply with all study procedures.
* Stated availability for the duration of the study.
* Ability to identify members of their social network who may benefit from receiving an HIVST kit and PrEP information.
* Currently prescribed PrEP by RAPID clinics, including those initiating PrEP on the same day as study enrollment.

Inclusion Criteria for Peers (Alters):

- Provision of electronic informed consent prior to completion of the Quick Response (QR)-linked survey instruments.

Exclusion Criteria for PrEP Clients (Egos):

* Inability or refusal to provide informed consent (e.g., cognitive impairment).
* Unable or unwilling to comply with study procedures per study investigator
* Inability to identify members of their social network who may benefit from receiving an HIVST kit and PrEP information.
* Aged 17 years or younger.

Exclusion Criteria for Peers (Alters):

* Failure to provide electronic informed consent prior to starting QR-linked Alter survey tools.
* Age 17 years or younger.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of Alter participants per ego who use the HIV self-test kit | Up to 6 months
  Number of Alter participants per ego who use an HIV self-test kit, indicated by completion of the Post-Test Survey.
Number of Alter participants per ego using an HIV self-test who meet criteria for PrEP | Up to 6 months
  Number of Alter participants per ego using an HIV self-test who meet criteria for PrEP

SECONDARY OUTCOMES:
Number of Alters per ego initiating PrEP | Up to 6 months
  Number of Alters per ego initiating PrEP
Alters' self-reported PrEP knowledge as indicated by the Post-Test Survey. | Up to 6 months
  Scores on Post-Test Survey range from 0-100. Higher scores indicate higher PrEP knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Dobleck-Lewis, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No